CLINICAL TRIAL: NCT00294034
Title: VIBRANT Registry: Value of Information Based From Pacemaker Recordings and New Technologies
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry); Medtronic BRC (Industry)
Other Study IDs: 197
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Pacemaker; Bradycardia
Keywords: Registry; Pacemaker; Diagnostics
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Pacemaker

SUMMARY:
The purpose of this study is to collect data from pacemakers and determine how this information is used by physicians to care for their patients with pacemakers.

DETAILED DESCRIPTION:
The purpose of this registry is to gain a better understanding of how diagnostic capabilities in four Vitatron pacemakers (Selection AFm, Clarity, C-Series, and T-Series) are being utilized for the clinical management of a general pacing population. Pacemaker information and health status is collected from all patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

• Class I or Class II indication for dual chamber pacing

Exclusion Criteria:

* Has an ICD or is a known candidate for an ICD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 950
Dates: Start 2002-10; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Jaffe, MD, Principal Investigator — Onondaga Hill Cardiovascular Group; Luis Caceres, MD, Principal Investigator — Prairie Cardiovascular Consultants
Locations (27):
- United States (27):
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Fort Lauderdale, Florida
  - Largo, Florida
  - Ormond Beach, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Hyannis, Massachusetts
  - Lansing, Michigan
  - Bay Shore, New York
  - Syracuse, New York
  - Bismarck, North Dakota
  - Barberton, Ohio
  - Cincinnati, Ohio
  - Marion, Ohio
  - Massillon, Ohio
  - Middletown, Ohio
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Arlington, Texas
  - Austin, Texas
  - Beaumont, Texas
  - McKinney, Texas
  - Waukesha, Wisconsin